CLINICAL TRIAL: NCT05464862
Title: The Effect of the Popliteal Plexus Block on the Motor Function of the Leg - a Randomized, Controlled, Blinded Study in Volunteers
Brief Title: The Effect of PPB Using 10, 20 and 30 ml of Lidocaine, Study on Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charlotte Runge (Other)
Collaborators: Danish Society of Anesthesiology and Intensive Care Medicine (Unknown); University of Aarhus (Other); The Danish Rheumatism Association (Other)
Responsible Party: Sponsor-Investigator, Charlotte Runge, Medical Doctor, Specialist in Anesthesiology, PhD, Clinical Associate Professor, Regionshospitalet Silkeborg
Organization: Regionshospitalet Silkeborg (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-501206-35-00
Record Dates: First submitted 2022-07-05; First posted 2022-07-19 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Knee Arthritis; Anesthesia, Local; Post Surgical Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A randomization list is computed by the REDCap administrator from Aarhus University and imported in REDCap.The anesthesiologist and the assistant performing all the nerve blocks, are the only one with access to REDCaps randomization module, where the randomization procedure is made prior to the nerve block procedure.
  The randomization list will assign each volunteer to one of six combinations, deciding which type of peripheral nerve block is used for each their leg. One leg equal one observation. The combinations ensure that observations are obtained in even numbers from right and left legs and that the total dose of perineural used lidocaine does not exceed 400 mg per volunteer.
  Groups name, type of peripheral nerve block, study medication dosage and number of legs in the group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study is an assessor- and volunteer-blinded randomized study. As different volumes are used for the nerve blocks, the anesthesiologist and an assistant performing the nerve blocks will not be blinded, and therefore have no further contact with the volunteers after the nerve block performance and will not contribute with the data collection or statistical analysis. The nerve block procedure and assessments will take place in different rooms; hence the data collecting assessors will not be present during block performance.To ensure blinding of the volunteer, a draping will hinder the volunteer from observing which volume of lidocaine that is administered during block performance.Group A, B and C are blinded until the data analysis is finished. Group FNB of SNB are unblinded and works as active comparatives for model control, in order to establish reference points for when a nerve is considered affected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group A (Experimental): Popliteal Plexus Block given with 10 ml of Lidocaine Hydrochloride 10 mg/ml
  Interventions: Drug: Popliteal Plexus Block with 10 ml
- Groups B (Experimental): Popliteal Plexus Block given with 20 ml of Lidocaine Hydrochloride 10 mg/ml
  Interventions: Drug: Popliteal Plexus Block with 20 ml
- Group C (Experimental): Popliteal Plexus Block given with 30 ml of Lidocaine Hydrochloride 10 mg/ml
  Interventions: Drug: Popliteal Plexus Block with 30 ml
- Group FNB (Active Comparator): Femoral Nerve Block given with 20 ml of Lidocaine Hydrochloride 10 mg/ml
  Interventions: Drug: Femoral Nerve Block
- Groups SNB (Active Comparator): Sciatic Nerve Block given with 20 ml og Lidocaine Hydrochloride 10 mg/ml
  Interventions: Drug: Sciatic Nerve Block

INTERVENTIONS:
Drug: Popliteal Plexus Block with 10 ml — Ultrasound-guided Popliteal Plexus Block using 10 ml of of Lidocaine Hydrochloride 10 mg/ml
  Arms: Group A
Drug: Popliteal Plexus Block with 20 ml — Ultrasound-guided Popliteal Plexus Block using 20 ml of of Lidocaine Hydrochloride 10 mg/ml
  Arms: Groups B
Drug: Popliteal Plexus Block with 30 ml — Ultrasound-guided Popliteal Plexus Block using 30 ml of of Lidocaine Hydrochloride 10 mg/ml
  Arms: Group C
Drug: Femoral Nerve Block — Ultrasound-guided Femoral Nerve Block using 20 ml of of Lidocaine Hydrochloride 10 mg/ml. Is used to find cut-off values that define affection of the femoral nerve.
  Arms: Group FNB
Drug: Sciatic Nerve Block — Ultrasound-guided Sciatic Nerve Block using 20 ml of of Lidocaine Hydrochloride 10 mg/ml. Is used to find cut-off values that define affection of the sciatic nerve.
  Arms: Groups SNB

SUMMARY:
The aim of this study is to evaluate the Popliteal Plexus Block (PPB) effect on motor nerve branches of the sciatic and femoral nerve, when using different volumes of local anesthetics for PPB.

The hypothesis is that increasing the volume of anesthetics used for PPB will spread to the sciatic nerve leading to a reduced muscle strength in the lower leg and decreased nerve conduction velocity in the nerve to gastrocnemius muscle (the tibial nerve) and the nerve to anterior tibial muscle (the deep fibular nerve).

The effects will be evaluated by maximum voluntary isometric contraction (MVIC) of the lower leg muscles and by recordings of the compound muscle action potential (cMAP) of the gastrocnemius and tibialis anterior muscles - a motor nerve conduction study.

In addition, evaluation of PPBs effect on the femoral nerve is done by MVIC of the quadriceps femoris muscle, cMAP of the vastus medialis and vastus lateralis muscles and by a sensory nerve conduction study of the saphenous nerve.

DETAILED DESCRIPTION:
A total number of 40 volunteers will be enrolled in the study. Each volunteer will receive two peripheral nerve blocks (one in each leg) on the day of participation. This will result in 80 peripheral nerve blocks. The types of nerve blocks given to each leg on each volunteer will depend on randomization.

The 80 nerve blocks are divided into five groups specified by type of nerve block, volume of anesthetic used, and respective numbers of legs used in the group. The groups and specifications are listed here:

Groups name, type of peripheral nerve block, study medication dosage and number of legs in the group:

* Group A: PPB with 10 ml of lidocaine 1%, 20 legs.
* Group B: PPB with 20 ml of lidocaine 1%, 20 legs.
* Group C: PPB with 30 ml of lidocaine 1%, 20 legs.
* Group FNB: FNB with 20 ml of lidocaine 1%, 10 legs.
* Group SNB: SNB with 20 ml of lidocaine 1%, 10 legs.

Group FNB of SNB are performed unblinded and works as active comparatives for model control, in order to establish reference points for when a nerve is considered affected.

Prior to nerve block procedure , pre block assessments are obtained in the following order:

* Sensory test of the saphenous nerve.
* MVIC by ankle plantarflexion.
* MVIC by ankle dorsiflexion.
* MVIC by knee extension.
* Compound muscle action potential (cMAP) recordings in the following order:

  * Nerve to vastus medialis muscle
  * Nerve to vastus lateralis muscle
  * Nerve to tibialis anterior muscle
  * Nerve to gastrocnemius muscle

    60 minutes after the block performance, post block assessments are done. Values are obtained in the same order as for the pre block assessments.

A peripheral intravenous line is inserted prior to the procedure of the peripheral nerve block is performed. At the discretion of the anesthetist, up to 20 mg Propofol IV may be provided to ease the patient during the nerve block procedure. The volunteer is monitored with continuous electrocardiography and pulse oximetry for the first 30 minutes after block performance and clinically hereafter. Final check by an investigator to ensure the volunteer is ready to go home. If the muscle strength is reduced, the volunteer will not be sent home before the ability to walk safely with crutches is ensured.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* Ability to give their written informed consent to participating in the study after having fully understood the contents of the study

Exclusion Criteria:

* Subjects who cannot cooperate with the study.
* Subjects who cannot understand or speak Danish.
* Subjects with allergy to the medicines used in the study.
* Subjects suffering from alcohol and/or drug abuse - based on the investigator's opinion.
* Pathology or previous major surgery to the lower limb.
* Intake of any analgesics 24 hours prior to baseline measurements.
* BMI > 35
* Active signs of infection in the cutaneous area of injection
* Subjects diagnosed with epilepsy, neurologic diseases, severe hypoxia or respiratory depression, hypovolemia, shock, bradycardia or Wolff-Parkinson-Whites syndrome
* Subjects with a positive pregnancy test**
* Subjects diagnosed with cardiovascular disease or heart failure
* Subjects diagnosed with partial or complete cardiac block
* Subjects in daily treatment with class III antiarrhythmics (e.g. amiodarone)
* Subjects in daily treatment with drugs that are structurally related to local analgesics or class IB antiarrhythmics
* Subjects diagnosed with severe liver disease or reduced kidney function

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
MVIC (Maximum Voluntary Isometric Contraction) ankle plantarflexion | Measured pre block and at 45 minutes post block
  Difference between group A, B and C in post block MVIC by ankle plantarflexion, expressed as percentage change of the pre block value. MVIC is measured using a handheld dynamometer.
MVIC ankle dorsiflexion | Measured pre block and at 45 minutes post block
  Difference between group A, B and C in post block MVIC by ankle dorsiflexion, expressed as a percentage change of the pre block value. MVIC is measured using a handheld dynamometer.

SECONDARY OUTCOMES:
MVIC knee extension | Measured pre block and at 45 minutes post block
  Difference between group A, B and C in post block MVIC by knee extension, expressed as a percentage change of the pre block value. MVIC is measured using a handheld dynamometer.
cMAP (compoud motor action potention) gatrocnemius | Measured pre block and at 45 minutes post block
  Difference between group A, B and C, in the number of volunteers with affected cMAP of the gastrocnemius muscle, defined as sufficient change from pre block to post block. Cut-off value for sufficient change is determined by SNB group. cMAP is recorded using a motor nerve conduction study.
cMAP tibialis anterior | Measured pre block and at 45 minutes post block
  Difference between group A, B and C, in the number of volunteers with affected cMAP of the tibialis anterior muscle, defined as sufficient change from pre block to post block. Cut-off value for sufficient change is determined by SNB group. cMAP is recorded using a motor nerve conduction study.
cMAP vastus medialis | Measured pre block and at 45 minutes post block
  Difference between group A, B and C, in the number of volunteers with affected cMAP of the vastus medialis muscle, defined as sufficient change from pre block to post block. Cut-off value for sufficient change is determined by FNB group. cMAP is recorded using a motor nerve conduction study.
cMAP vastus lateralis | Measured pre block and at 45 minutes post block
  Difference between group A, B and C, in the number of volunteers with affected cMAP of the vastus lateralis muscle, defined as sufficient change from pre block to post block. Cut-off value for sufficient change is determined by FNB group. cMAP is recorded using a motor nerve conduction study.
Saphenus senory test | Measured pre block and at 45 minutes post block
  Difference between group A, B and C in the number of volunteers with an affected sensory of the saphenous nerve, defined as change, from pre block to post block, in the volunteers ability to discriminate cold in the cutaneous area innervated by the medial crural cutaneous branches of saphenous nerve.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Sørensen, MD, Principal Investigator — Aarhus Universitet (Aarhus)
Locations (1):
- Elective Surgery Center at Silkeborg Regional Hospital, Silkeborg, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after acceåtance from The Danish Data Protection Agency
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of the study analysis
Access Criteria: Permission by investigators

REFERENCES:
- [Derived] Sorensen JK, Grevstad U, Qerama E, Bruun LS, Nikolajsen L, Runge C. Effect of local anesthetic volume for popliteal plexus block on motor nerve conduction and muscle function in the leg: a randomized clinical trial in healthy volunteers. Reg Anesth Pain Med. 2025 Apr 3:rapm-2025-106557. doi: 10.1136/rapm-2025-106557. Online ahead of print. PMID 40185510